CLINICAL TRIAL: NCT03563599
Title: An Open-label Randomized Study to Evaluate the Early Bactericidal Activity, Safety, Tolerability, and Pharmacokinetics of Multiple Oral Doses of Telacebec (Q203) in Treatment-naïve Patients With Newly Diagnosed Drug-sensitive Sputum Smear-positive Pulmonary Tuberculosis
Brief Title: A Phase 2 Study to Evaluate Early Bactericidal Activity, Safety, Tolerability, and Pharmacokinetics of Multiple Oral Doses of Telacebec (Q203)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Qurient Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Q203-TB-P2-ZA001
Record Dates: First submitted 2018-06-09; First posted 2018-06-20 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Treatment-naïve, Sputum Smear-positive Patients With Drug-sensitive Pulmonary TB
MeSH Terms: interventions — telacebec

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Telacebec (Q203) tablet (Experimental)
  Interventions: Drug: Telacebec (Q203)
- Rifafour e-275 (Active Comparator)
  Interventions: Drug: Rifafour e-275

INTERVENTIONS:
Drug: Telacebec (Q203) — High, Mid, Low dose of telacebec
  Arms: Telacebec (Q203) tablet
Drug: Rifafour e-275 — RHZE (R=rifampicin: H=isoniazid: Z=pyrazinamide: E=ethambutol)
  Arms: Rifafour e-275

SUMMARY:
This is a Phase IIa, open-label, randomized study in treatment-naïve, sputum smear-positive patients with drug-sensitive pulmonary TB to assess the early bactericidal activity of telacebec (Q203).

ELIGIBILITY:
Inclusion Criteria:

1. A new episode of pulmonary TB determined by testing at the study appointed laboratory: Mycobacterium tuberculosis positive and rifampicin and isoniazid sensitive on a rapid molecular test
2. A chest X-ray taken no more than 14 days before Screening which in the opinion of the Investigator is consistent with TB
3. Sputum smear positive on direct microscopy for acid-fast bacilli on at least 1 pre-treatment sputum sample
4. Ability to produce an adequate volume of sputum as determined by an approximately 16-hour overnight sample collection
5. Be of non-childbearing potential or using effective methods of birth control, as defined in the protocol

Exclusion Criteria:

1. The patient is mentally or legally incapacitated at Screening
2. Any condition or circumstance, in the opinion of the Investigator, which may make the patient unlikely to complete the study or comply with study procedures and requirements, or may pose a risk to the patient's safety
3. Clinically significant evidence of extra-thoracic TB (miliary TB, abdominal TB, urogenital TB, osteoarthritic TB, TB meningitis), as judged by the Investigator
4. The patient has been infected with hepatitis B or C virus as confirmed by tests for hepatitis B core antibodies, hepatitis B surface antigens, and the hepatitis C virus antibodies
5. The patient with history of allergic reaction to isoniazid, rifampicin, pyrazinamide, ethambutol or related substances (eg, tosylate), as confirmed by the clinical judgement of the Investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-07-23 (Actual); Primary Completion 2019-09-09 (Actual); Study Completion 2019-09-09 (Actual)

PRIMARY OUTCOMES:
The EBA (early bactericidal activity) of telacebec (Q203) | Days 0 to 14 post dose
  The EBA determined by the rate of change in the time to positivity (TTP) in sputum over the periods Days 0 to 14

CONTACTS AND LOCATIONS:
Locations (2):
- South Africa (2):
  - TASK Applied Science, Cape Town
  - UCT Lung Institute, Cape Town

REFERENCES:
- [Derived] Janssen S, Upton C, de Jager VR, van Niekerk C, Dawson R, Hutchings J, Kim J, Choi J, Nam K, Sun E, Diacon AH. Telacebec, a Potent Agent in the Fight against Tuberculosis: Findings from a Randomized, Phase 2 Clinical Trial and Beyond. Am J Respir Crit Care Med. 2025 Aug;211(8):1504-1512. doi: 10.1164/rccm.202408-1632OC. PMID 40116781